CLINICAL TRIAL: NCT06594874
Title: A Phase Ib Study Evaluating the Safety, Tolerability , Pharmacokinetics and Activity of HS-10370 in Addition to Other Anti-cancer Therapies in Participants with KRAS G12C Mutation Advanced Solid Tumors
Brief Title: A Phase Ib Study of HS-10370 in Addition to Other Anti-cancer Therapies in Participants with KRAS G12C Mutation Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10370-102
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer; Advanced Solid Tumors
Keywords: KRAS G12C; Non-Small Cell Lung Cancer; Metastatic Solid Tumor; Adebrelimab; Carboplatin; Pemetrexed; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm A: HS-10370 dose 1 + Adebrelimab (Experimental): Participants will receive HS-10370 dose 1 administered orally plus Adebrelimab given as a 20 mg/kg intravenous infusion(IV) once every 21-day cycle up to a total of 35 cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: HS-10370; Drug: Adebrelimab
- Arm B: HS-10370 dose 2 + Adebrelimab (Experimental): Participants will receive HS-10370 dose 2 administered orally plus Adebrelimab given as a 20 mg/kg intravenous infusion(IV) once every 21-day cycle up to a total of 35 cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: HS-10370; Drug: Adebrelimab
- Arm C: HS-10370+ Adebrelimab + Pemetrexed and Platinum (Experimental): Participants will receive HS-10370 administered orally in plus with Adebrelimab, pemetrexed, and platinum (cisplatin or carboplatin) administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met
  Interventions: Drug: HS-10370; Drug: Adebrelimab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Arm D: HS-10370+ Adebrelimab + Pemetrexed (Experimental): Participants will receive HS-10370 administered orally in plus with Adebrelimab and pemetrexed administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: HS-10370; Drug: Adebrelimab; Drug: Pemetrexed
- Arm E: HS-10370+ Pemetrexed and Platinum (Experimental): Participants will receive HS-10370 administered orally in plus with pemetrexed and platinum (cisplatin or carboplatin) administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: HS-10370; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: HS-10370 — HS-10370 administered orally every day
Drug: Adebrelimab — Administered intravenously every 21 days; dose by label.
  Arms: Arm A: HS-10370 dose 1 + Adebrelimab; Arm B: HS-10370 dose 2 + Adebrelimab; Arm C: HS-10370+ Adebrelimab + Pemetrexed and Platinum; Arm D: HS-10370+ Adebrelimab + Pemetrexed
Drug: Cisplatin — Administered intravenously every 21 days; dose by label.
  Arms: Arm C: HS-10370+ Adebrelimab + Pemetrexed and Platinum; Arm E: HS-10370+ Pemetrexed and Platinum
Drug: Carboplatin — Administered intravenously every 21 days; dose by label.
  Arms: Arm C: HS-10370+ Adebrelimab + Pemetrexed and Platinum; Arm E: HS-10370+ Pemetrexed and Platinum
Drug: Pemetrexed — Administered intravenously every 21 days; dose by label.
  Arms: Arm C: HS-10370+ Adebrelimab + Pemetrexed and Platinum; Arm D: HS-10370+ Adebrelimab + Pemetrexed; Arm E: HS-10370+ Pemetrexed and Platinum

SUMMARY:
This is a Phase Ib study that will evaluate the Safety, Tolerability , Pharmacokinetics and Activity of HS-10370 in Combination With Other Anti-cancer Therapies in patients with KRAS G12C mutation advanced or metastatic solid tumors, especially in non-Small cell lung cancer (NSCLC) .

ELIGIBILITY:
Inclusion Criteria:

* Men or women greater than or equal to 18 years
* At least one measurable lesion in accordance with RECIST 1.1
* Must have an ECOG performance status of 0 or 1.
* Histologically or cytologically confirmed NSCLC with Stage IIIB-IIIC or Stage IV disease, not suitable for curative intent radical surgery or radiation therapy.
* Documentation of the presence of a KRAS G12C mutation
* Must provide tumor tissue sample
* No history of systemic anticancer therapy in metastatic/non-curable settings
* Estimated life expectancy ≥12 weeks.
* Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 6 months after the last dose.
* Females must have the evidence of non-childbearing potential; Likewise, men also consent to use adequate contraceptive method within the same time limit.
* Signed and dated Informed Consent Form.
* The subjects are able to comply with the process of the protocol.

Exclusion Criteria:

* Treatment with any of the following:

  1. Previous or current treatment with other KRAS G12C inhibitors
  2. Any cytotoxic chemotherapy, anticancer Chinese medicine and targeted small molecule inhibitors within 14 days of the first dose of study treatment; Any investigational agents and large molecule antibodies within 28 days of the first dose of study treatment.
  3. Local radiotherapy within 2 weeks prior to the first dose of study drug, more than 30% of bone marrow irradiation or large-area radiotherapy within 4 weeks before the first dose of study drug.
  4. Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose
* Active brain metastases.
* Patients with uncontrolled pleural, ascites or pericardial effusion
* Spinal cord compression
* Presence of Grade ≥ 2 toxicities due to prior anti-tumor therapy.
* Subjects with tumors known to harbor molecular alterations for which targeted therapy is locally approved, except for KRAS G12C.
* History of other primary malignancies.
* Inadequate bone marrow reserve or organ functions.
* Abnormal cardiac examination results.
* Severe, uncontrolled or active cardiovascular disorders.
* Diabetes ketoacidosis or hyperglycemia hyperosmolality
* Uncontrolled hypertension.
* Severe bleeding symptoms or bleeding tendencies.
* Severe arteriovenous thrombosis occurred
* Serious infection.
* Continuous use of glucocorticoids
* Active infectious diseases.
* Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow oral medications
* Hepatic encephalopathy, hepatorenal syndrome, or ≥ Child Pugh B-grade cirrhosis.
* Interstitial lung disease (ILD).
* Serious neurological or mental disorders.
* Active autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Event(s) (AEs) | From Cycle 1 Day 1 to first documented progression of disease or death from any cause, approximately 2 years.
  An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment. Severity is determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From Cycle 1 Day 1 (C1D1) to disease progression or death, approximately 2 years.
  Percentage of Participants who Achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR).ORR by the Investigator According to RECIST v1.1
Disease Control Rate (DCR) | From C1D1 to disease progression or death, approximately 2 years.
  Percentage of Participants who Achieve a BOR of CR, PR, or Stable Disease (SD).DCR by the Investigator According to RECIST v1.1
Time to Response (TTR) | Time from C1D1 until the date that measurement criteria for CR or PR (whichever is first recorded) are first met, approximately 2 years.
  TTR by the Investigator According to RECIST v1.1
Duration of Response (DOR) | Date of first evidence of CR or PR to date of disease progression or death from any cause, approximately 2 years.
  DOR by the Investigator According to RECIST v1.1
Progression-Free Survival (PFS) | Date of first evidence of CR or PR to date of disease progression or death from any cause, approximately 2 years.
  PFS by the Investigator According to RECIST v1.1
Overall survival (OS) | C1D1 to date of death from any cause, approximately 5 years.
  Defined as the time from C1D1 to death from any cause
Plasma Concentrations of HS-10370 | C1D1 to date of death from any cause. Various timepoints from Cycle 1 Day 1 through study treatment discontinuation, approximately 2 years.
  Defined as the time from C1D1 to death from any cause
Maximum plasma concentration (Cmax) | C1D1 to date of death from any cause, approximately 2 years. Various timepoints from Cycle 1 Day 1 through study treatment discontinuation.
  Cmax is defined as maximum observed serum concentration obtained directly from the observed concentration-time data.
Time of maximum concentration (Tmax) | C1D1 to date of death from any cause, approximately 2 years. Various timepoints from Cycle 1 Day 1 through study treatment discontinuation
  Tmax is defined as the time required for a drug to reach peak concentration in plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Tong Ji Medical College, HuaZhong University of Science and Technology, Wuhan, Hubei, China